CLINICAL TRIAL: NCT06226571
Title: A Phase 1, Open-label, Dose-escalation, and Dose-expansion Study to Evaluate Safety, Tolerability, and Clinical Activity of SNDX-5613 in Combination With Intensive Chemotherapy in Participants With Newly Diagnosed Acute Myeloid Leukemias Harboring Alterations in Lysine-specific Methyltransferase 2A (KMT2A/MLL), Nucleophosmin 1 (NPM1), and Nucleoporin 98 (NUP98) Genes
Brief Title: A Study of SNDX-5613 in Combination With Intensive Chemotherapy in Participants With Acute Myeloid Leukemias
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-5613-0708; 2024-514531-18-00 (EU CTIS Number)
Expanded Access: NCT05918913 (No longer available)
Record Dates: First submitted 2024-01-12; First posted 2024-01-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemias
Keywords: SNDX-5613; Lysine-specific Methyltransferase 2A; KMT2A/MLL; Nucleophosmin 1; NPM1; Nucleoporin 98; NUP98; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SNDX-5613 (Experimental): Dose Escalation:
  * Induction: Sequential cohorts of escalating dose levels of SNDX-5613 with chemotherapy regimen.
  * Consolidation: Cohorts will receive high-dose cytarabine (HiDAC) chemotherapy followed by SNDX-5613.
  * Maintenance Monotherapy: Cohorts will receive SNDX-5613.
  Dose Expansion:
  * Induction: SNDX-5613 at tolerated dose level with chemotherapy regimen.
  * Consolidation: Cohorts will receive SNDX-5613 with chemotherapy regimen and HiDAC.
  * Maintenance Monotherapy: Cohorts will receive SNDX-5613.
  Interventions: Drug: SNDX-5613; Drug: Chemotherapy Regimen; Drug: HiDAC

INTERVENTIONS:
Drug: SNDX-5613 — Participants will receive SNDX-5613 orally during Induction, Consolidation, and Maintenance until meeting criteria for discontinuation.
Drug: Chemotherapy Regimen — Induction: Participants will receive an intravenous (IV), 2-drug combination of cytarabine and either daunorubicin or idarubicin.
Drug: HiDAC — Consolidation: Participants will receive HiDAC IV.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and clinical activity of SNDX-5613 in combination with intensive chemotherapy in participants with newly diagnosed acute myeloid leukemia (AML) harboring alterations in KMT2A, NPM1, or NUP98 genes.

DETAILED DESCRIPTION:
The Dose Escalation portion of this study will identify the maximum tolerated dose, or if different, the recommended Phase 2 dose of SNDX-5613 to be used in combination with intensive chemotherapy and in maintenance monotherapy following intensive chemotherapy in participants with newly diagnosed AML harboring alterations in KMT2A, NPM1, or NUP98 genes.

In the Dose Expansion portion of the study, safety and preliminary efficacy of SNDX-5613 may be explored in expansion cohorts at tolerated dose levels.

In both Dose Escalation and Dose Expansion, the treatment period will consist of an induction phase (up to 2 cycles), a consolidation phase (up to 4 cycles and could include hematopoietic stem cell transplant for participants who are transplant eligible and have an available donor), and a maintenance monotherapy phase with SNDX-5613. The cycle duration will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Established, pathologically confirmed diagnosis of AML by World Health Organization 2022 criteria.
* Previously untreated AML and eligible to receive intensive chemotherapy.
* KMT2Ar, NPM1c, or NUP98r mutations identified by local laboratory prior to the first dose of SNDX-5613.
* Eastern Cooperative Oncology Group performance status ≤2 and ≤1 if >65 years old .
* Adequate liver, kidney, and cardiac function.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia.
* Clinically active central nervous system leukemia (blasts detected in cerebrospinal fluid, radiographic or clinical signs and symptoms).
* Fridericia's corrected QT interval (QTcF) >450 milliseconds (average of triplicate), diagnosis or suspicion of Long QT syndrome or family history of Long QT syndrome.
* Any gastrointestinal issue of the upper gastrointestinal tract that might affect oral drug absorption or ingestion.
* Cirrhosis with a Child-Pugh score of B or C.
* Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
* Hepatitis B, Hepatitis C, or HIV-positive with detectable viral load.
* Documented active, uncontrolled infection.
* Uncontrolled disseminated intravascular coagulation.
* Lactating/breast feeding or pregnant.
* Use of prohibited concomitant chemotherapy, radiation therapy, or immunotherapy.
* Use of strong CYP3A4 inducers or inhibitors (except for Itraconazole, Ketoconazole, Posaconazole, or Voriconazole).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Number of Participants with Dose-limiting Toxicities | Up to Day 42
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 through 30 days after final dose (up to approximately 3 years)

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of SNDX-5613 and Relevant Metabolites | Predose through Day 15
Area Under the Plasma Concentration Versus Time Curve From Time 0 to t (AUC0-t) of SNDX-5613 and Relevant Metabolites | Predose through Day 15

CONTACTS AND LOCATIONS:
Locations (43):
- United States (25):
  - UCLA Medical Hematology, Burbank, California
  - City of Hope Medical Center, Duarte, California
  - AdventHealth Blood & Marrow Transplant Center, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Institution name: Northwell Health-Brany, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - East Carolina University, Greenville, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University- Center for Hematologic Malignancies, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center (HCC), Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - LDS Hospital - Intermountain Healthcare, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia
- Australia (5):
  - Northern Hospital, Victoria, Epping, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - The Alfred Hospital, Victoria, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
- Gordon and Leslie Diamond Health Care Center, Vancouver, British Columbia, Canada
- University Medical Center Utrecht, Utrecht, Netherlands
- Spain (9):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario De Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Universitat de Valencia, Valencia
- United Kingdom (2):
  - Hammersmith Hospital, London, London, City of
  - The Royal Marsden NHS, Sutton

IPD SHARING:
Plan to Share IPD: No